CLINICAL TRIAL: NCT06966401
Title: A Long-Term, Open-Label Study to Assess the Safety and Tolerability of NBI-1065845 as Adjunctive Treatment in Subjects With Major Depressive Disorder (MDD)
Brief Title: Long-Term Study to Assess the Safety and Tolerability of NBI-1065845 as an Adjunctive Treatment in Participants With Major Depressive Disorder (MDD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-1065845-MDD3028; 2024-519423-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-30; First posted 2025-05-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression; Major Depressive Disorder; NBI-1065845; TAK-653
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBI-1065845 (Experimental): NBI-1065845 administered orally once a day.
  Interventions: Drug: NBI-1065845

INTERVENTIONS:
Drug: NBI-1065845 — NBI-1065845 tablets
  Other Names: TAK-653

SUMMARY:
This study will evaluate the long-term safety and tolerability of NBI-1065845 as an adjunctive treatment in participants with MDD.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of recurrent MDD (moderate or severe) or persistent depressive disorder.
* Participant has had an inadequate response to oral antidepressant treatments in the current episode of depression.
* Participant must have been taking oral antidepressants for at least 8 weeks prior to screening.
* Willing and able to comply with all study procedures and restrictions in the opinion of the investigator.

Key Exclusion Criteria:

* A current or prior psychiatric disorder diagnosis in the last 1 year that was the primary focus of treatment other than MDD.
* Are considered by the investigator to be at imminent risk of suicide or injury to self or others.

Other protocol defined inclusion and exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Baseline through Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (18):
- United States (18):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, Pico Rivera, California
  - Neurocrine Clinical Site, Upland, California
  - Neurocrine Clinical Site, Hollywood, Florida
  - Neurocrine Clinical Site, Maitland, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Watertown, Massachusetts
  - Neurocrine Clinical Site, Saint Charles, Missouri
  - Neurocrine Clinical Site, Mount Kisco, New York
  - Neurocrine Clinical Site, The Bronx, New York
  - Neurocrine Clinical Site, Avon Lake, Ohio
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Richmond, Texas
  - Neurocrine Clinical Site, The Woodlands, Texas
  - Neurocrine Clinical Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No